CLINICAL TRIAL: NCT01951703
Title: Clinical Investigation of Senofilcon A Manufactured Using an Alternate Hydration Process
Brief Title: Senofilcon A Investigational Manufacturing Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CR-5509
Record Dates: First submitted 2013-09-23; First posted 2013-09-27 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-04

CONDITIONS: Visual Acuity; Comfort; Overall Vision

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control, senofilcon A (Active Comparator): Subjects received Control lens, senofilcon A during the first two weeks of the study then Test lens, senofilcon A in the last two weeks of the study.
  Interventions: Device: senofilcon A
- Test, senofilcon A (Experimental): Subjects received Test lens, senofilcon A during the first two weeks of the study then Control lens, senofilcon A in the last two weeks of the study.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A — Control, senfilcon A
  Arms: Control, senofilcon A
Device: senofilcon A — Test, senofilcon A
  Arms: Test, senofilcon A

SUMMARY:
To evaluate the impact of a new contact lens hydration process

DETAILED DESCRIPTION:
To evaluate the impact on clinical performance of senofilcon A lenses manufactured using an alternate hydration process and compare the performance with senofilcon A lenses manufactured using the current process.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be at least 18 and not more than 70 years of age.
* The subject's refractive cylinder must be < 0.75D in each eye.
* The subject must have best corrected visual acuity of 20/25 or better in each eye.
* The subject must demonstrate adequate mobility and 20/30 vision OD and OS with the study contact lenses.
* The subject must be a habitual and adapted wearer of ACUVUE® OASYS® Brand contact lens in both eyes.
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).
* The subject's required spherical contact lens prescription must be in the range of -0.50 to -9.00D in each eye.

Exclusion Criteria:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
* Any systemic disease, autoimmune disease, or use of medication, that may interfere with contact lens wear.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any known hypersensitivity or allergic reaction to OPTI-FREE® PureMoist® Contact Lens Solution.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Monovision or multi-focal contact lens correction.
* Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
* History of binocular vision abnormality or strabismus.
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self report).
* Suspicion of or recent history of alcohol or substance abuse.
* History of serious mental illness.
* History of seizures.
* Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pall, OD, Study Director — Johnson & Johnson Vision Care
Locations (4):
- United States (4):
  - Jacksonville, Florida
  - Bloomington, Illinois
  - Pittsburg, Kansas
  - Warwick, Rhode Island

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 136 subjects were enrolled in the study; 9 subjects did not meet the inclusion and exclusion criteria and not randomized. Of the 127 randomized subjects, 6 were prematurely discontinued from the study and 2 were excluded from the analysis due to major protocol deviations.
Groups:
- Control/Test: Subjects that received Control lens, senofilcon A for the first two weeks and then received Test lens senofilcon A in the last two weeks of the study.
- Test/Control: Subjects that received Test lens, senofilcon A for the first two weeks and then received Control lens senofilcon A in the last two weeks of the study.
Period: First Intervention
Arm/Group | Control/Test | Test/Control
Started | 64 | 63
Completed | 61 | 62
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subject was not compliant | 1 | 1
Not completed — Physician Decision | 1 | 0
Period: Second Intervention
Arm/Group | Control/Test | Test/Control
Started | 61 | 62
Completed | 61 | 60
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Unsatisfactory Lens fitting | 0 | 1

BASELINE CHARACTERISTICS:
Population: This includes all randomized subjects
Groups:
- Control/Test: Subjects who received Control lens, senofilcon A for the first two weeks of the study and then received Test lens, senofilcon A in the last two weeks of the study.
- Test/Control: Subjects who received Test lens, senofilcon A for the first two weeks of the study and then received Control lens, senofilcon A in the last two weeks of the study.
- Total: Total of all reporting groups
Arm/Group | Control/Test | Test/Control | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 62 | 63 | 125
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (9.73) | 35.0 (9.63) | 35.2 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 102
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 61 | 56 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Comfort (Using CLUE )
Description: Contact Lens User Experience Comfort scores (CLUE) is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: 2 weeks
Population: Includes all subjects who completed all visits and did not have any major protocol deviation impacting the primary outcomes
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control, Senofilcon A: Subjects who received Control lens, senofilcon A in either the first two weeks or the last two weeks of the study.
- Test, Senofilcon A: Subject who received Test lens, senofilcon A in either the first two weeks or the last two weeks of the study.
Arm/Group | Control, Senofilcon A | Test, Senofilcon A
Number analyzed (Participants) | 119 | 119
units on a scale | 63.3 (24.85) | 65.0 (26.75)

2. Primary Outcome: Subjective Overall Vision (Using CLUE )
Description: Contact Lens User Experience Vision scores (CLUE) is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test, Senofilcon A: Subjects who received Test lens, senofilcon A in either the first two weeks or the last two weeks of the study.
Arm/Group | Control, Senofilcon A | Test, Senofilcon A
Number analyzed (Participants) | 119 | 119
units on a scale | 65.2 (20.75) | 65.2 (20.12)

ADVERSE EVENTS:
Groups:
- Test, Senofilcon A: Subjects who received Test lens senofilcon A in either the first two weeks or the last two weeks of the study,
Arm/Group | Control, Senofilcon A | Test, Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days